CLINICAL TRIAL: NCT01930591
Title: The Safety and Efficacy of Ticagrelor for Coronary Stenting Post Thrombolysis (SETFAST) Trial.
Brief Title: Ticagrelor for PCI Post Thrombolysis
Acronym: SETFAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Prairie Vascular Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 104
Record Dates: First submitted 2013-08-22; First posted 2013-08-29 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Acute Myocardial Infarction
Keywords: fibrinolytic therapy; stenting; platelet activity
MeSH Terms: interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel arm (Active Comparator): Clopidogrel 300 mg before PCI followed by 75 mg po OD
  Interventions: Drug: Clopidogrel
- Ticagrelor arm (Experimental): Ticagrelor 180 mg before PCI followed by 90 mg po BID
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — 180 mg bolus followed by 90 mg BID
  Other Names: Brilinta
  Arms: Ticagrelor arm
Drug: Clopidogrel — 300 mg bolus followed by 75 mg OD
  Other Names: Plavix
  Arms: Clopidogrel arm

SUMMARY:
Ticagrelor is a first line therapy along with aspirin for patients undergoing primary PCI for STEMI. However, many patients are still treated with fibrinolytic therapy and the safety and efficacy of Ticagrelor has not been investigated in this patients population. The present study is proposed to study the safety and efficacy of Ticagrelor in patients undergoing PCI post fibrinolytic therapy for STEMI.

DETAILED DESCRIPTION:
The newer antiplatelet agents such as Ticagrelor have demonstrated superiority to Clopidogrel in patients presenting with acute coronary syndrome (ACS). At present Ticagrelor remains a first line therapy as an adjunct to aspirin for patients undergoing primary PCI for STEMI for reducing major adverse events. However, the safety and efficacy of Ticagrelor has not been investigated in patients with STEMI post fibrinolysis. Ticagrelor results in significantly higher platelet inhibition than aspirin or clopidogrel and may expose patients to an increased risk of bleeding if administered post thrombolysis. However, fibrinolytic therapy itself results in a prothrombotic milieu with greater activation of platelets, a condition that can be balanced with addition of stronger antiplatelet agents. Similar concerns were initially reflected for clopidogrel as an adjunct to fibrinolytic therapy but were later proven to be unsubstantiated. In fact, adjunct administration of clopidogrel to fibrinolytic therapy reduces major adverse events as shown by multiple studies and has become the standard of care recommended by guidelines. The present study is proposed to study the safety and efficacy of Ticagrelor in patients undergoing PCI post fibrinolytic therapy for STEMI.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and over.
2. Planned PCI between 4-24 hours after administration of fibrinolytic therapy for STEMI.
3. Treatment with aspirin and clopidogrel as an adjunct to fibrinolytic therapy.
4. Informed written consent.

Exclusion Criteria:

1. Atrial fibrillation or need for systemic anticoagulation therapy.
2. Prior PCI or coronary artery bypass grafting during past 3 months.
3. Active bleeding or high risk of bleeding based upon clinical assessment.
4. Known severe liver or renal disease or patient requiring dialysis.
5. Concomitant oral or IV therapy with strong cytochrome (CYP3A) inhibitors which cannot be stopped.
6. Contraindication to ticagrelor or clopidogrel.
7. Planned surgery during the study period.
8. Any of the following in the absence of a functioning implanted pacemaker: sick sinus syndrome, 2nd or 3rd degree AVB, documented syncope of suspected bradycardic origin.
9. Known clinically important thrombocytopenia or anemia.
10. Known pregnancy or lactation.
11. Condition which may either put the patient at risk or influence the result of the study.
12. Previous randomization in this SETFAST study.
13. Participation in another clinical study with an investigational product or device study over the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-05; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Therapeutic platelet inhibition | 4 hours
  Therapeutic platelet inhibition as determined by VerifyNow assay (PRU value <208) at 4±1 hours post PCI

SECONDARY OUTCOMES:
Therapeutic platelet inhibition | 24 hours
  Therapeutic platelet inhibition (PRU value <208) at 24±4 hours post PCI.

OTHER OUTCOMES:
MACE | 24 hours or discharge
  MACE is a composite of death, re-infarction, stroke and bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Payam Dehghani, MD, Principal Investigator — Prairie Vascular Research Network, Regina, Saskatchewan; Asim Cheema, MD, Principal Investigator — St. Michael's Hospital, Toronto, Ontario
Locations (5):
- Canada (5):
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Prairie Vascular Research Inc. (PVRI), Regina General Hospital, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dehghani P, Lavoie A, Lavi S, Crawford JJ, Harenberg S, Zimmermann RH, Booker J, Kelly S, Cantor WJ, Mehta SR, Bagai A, Goodman SG, Cheema AN. Effects of ticagrelor versus clopidogrel on platelet function in fibrinolytic-treated STEMI patients undergoing early PCI. Am Heart J. 2017 Oct;192:105-112. doi: 10.1016/j.ahj.2017.07.013. Epub 2017 Jul 20. PMID 28938956